CLINICAL TRIAL: NCT03176238
Title: A Phase IIIb, Multi-center, Open-label Study of RAD001 in Combination With EXemestane in Post-menopausal Women With EStrogen Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: Study in Post-menopausal Women With Hormone Receptor Positive, HER2-negative Advanced Breast Cancer
Acronym: EVEREXES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001JIC06
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Post Menopausal Breast Cancer
Keywords: post menopausal; advanced breast cancer; metastatic breast cancer; everolimus; exemestane; mTor inhibitor; endocrine therapy; human epidermal growth factor; estrogen receptor positive; adult; CRAD001
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- everolimus + exemestane (Experimental): Everolimus (10 mg) and exemestane (25 mg) tablets taken orally in combination once daily
  Interventions: Drug: everolimus; Drug: exemestane

INTERVENTIONS:
Drug: everolimus — one 10 mg tablet or two 5 mg tablets of everolimus were administered orally once daily on a continuous dosing schedule starting on Day 1
  Other Names: RAD001
Drug: exemestane — 25 mg tablet was administered orally once daily on a continuous dosing schedule starting on Day 1

SUMMARY:
This international, multi-center, open-label, single-arm study evaluated the safety and tolerability profile of everolimus in post-menopausal women with HR positive, HER2 negative locally advanced or metastatic breast cancer after documented recurrence or progression following a non-steroidal aromatase inhibitors (NSAI) therapy in Novartis Oncology emergent growth market (EGM) countries.Data was presented by Asian countries vs Non-Asian countries to confirm no difference in safety and efficacy. Summary statistics were presented.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with metastatic, recurrent or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Histological or cytological confirmation of hormone-receptor positive (HR+) breast cancer.
* Disease refractory to non-steroidal aromatase inhibitors, defined as:
* Recurrence while on, or within 12 months (365 days) of completion of adjuvant therapy with letrozole or anastrozole, or
* Progression while on, or within one month (30 days) of completion of letrozole or anastrozole treatment for locally advanced or metastatic breast cancer (ABC).
* Radiological or objective evidence of recurrence or progression on or after the last systemic therapy prior to enrolment.
* Patients must have had:
* At least one lesion that could have been accurately measured in at least one dimension

  * 20 mm with conventional imaging techniques or ≥ 10 mm with spiral CT or MRI, or
* Bone lesions: lytic or mixed (lytic + blastic) in the absence of measurable disease as defined above.
* Adequate bone marrow, coagulation, liver and renal function.
* ECOG performance status ≤ 2.

Exclusion Criteria:

* Patients overexpressing HER2 by local laboratory testing (IHC 3+ staining or in situ hybridization positive). Patients with IHC 2+ must have a negative in situ hybridization test.
* Patients with only non-measurable lesions other than bone metastasis (e.g. pleural effusion, ascites).
* Patients with more than one prior chemotherapy line for ABC. A chemotherapy line is an anticancer regimen(s) that contained at least 1 cytotoxic chemotherapy agent, given for a minimum of 21 days.
* Previous treatment with mTOR inhibitors.
* Known hypersensitivity to mTOR inhibitors, e.g. Sirolimus (rapamycin).
* Patients with a known history of HIV seropositivity. Screening for HIV infection at baseline was not required.
* Patient who were being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A
* History of brain or other CNS metastases, including leptomeningeal metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- Australia (7):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Caringbah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Ringwood East, Victoria
  - Novartis Investigative Site, St Albans, Victoria
- India (4):
  - Novartis Investigative Site, Karamsad, Gujarat
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Cuttack, Odisha
- Indonesia (4):
  - Novartis Investigative Site, Bandung
  - Novartis Investigative Site, Jakarta
  - Novartis Investigative Site, Semarang
  - Novartis Investigative Site, Yogyakarta
- Novartis Investigative Site, Amman, Jordan
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur, MYS
  - Novartis Investigative Site, Kota Kinabalu, Sabah
- Morocco (2):
  - Novartis Investigative Site, Casablanca
  - Novartis Investigative Site, Rabat
- South Africa (3):
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Western Cape, Western Cape
- South Korea (8):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Jeollanam-do, Jeollanam-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Taiwan (5):
  - Novartis Investigative Site, Kaoshiung, Taiwan
  - Novartis Investigative Site, New Taipei City, TWN
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Novartis Investigative Site, Aryanah, Tunisia
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kartal
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred eleven participants were screened and 235 enrolled in Asian and non-Asian countries. Primary reason for discontinuation was presented.
Groups:
- Asian Everolimus + Exemestane: Everolimus (10 Mg) and exemestane (25 mg) tablets taken orally in combination once daily. Participants in Asian countries: Indonesia, India, Vietnam, Turkey, South Korea, Thailand, Malaysia, Taiwan or Jordan.
- Non-Asian Everolimus + Exemestane: Everolimus (10 mg) and exemestane (25 mg) tablets taken orally in combination once daily. Participants in Non-Asian countries: Australia, Morocco, South Africa or Tunisia.
Period: Overall Study
Arm/Group | Asian Everolimus + Exemestane | Non-Asian Everolimus + Exemestane
Started | 199 | 36
Completed | 0 | 0
Not Completed | 199 | 36
Not completed — Unacceptable AEs | 15 | 8
Not completed — Abnormal lab value(s) | 2 | 0
Not completed — Inter-current illness | 0 | 1
Not completed — Consent withdrawal | 14 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Death | 3 | 0
Not completed — Disease Progression | 133 | 22
Not completed — Tx duration completed per EAP | 0 | 1
Not completed — Patient is switched to commercial drug | 16 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Changes in the patient's condition | 2 | 1
Not completed — Everolimus dose interrupt > 4 wks | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asian Everolimus + Exemestane | Non-Asian Everolimus + Exemestane | Total
Number analyzed (Participants) | 199 | 36 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.00) | 60.8 (10.26) | 58.8 (10.05)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 199 | 36 | 235
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7 | 27 | 34
  Asian | 156 | 3 | 159
  Other | 36 | 6 | 42

OUTCOME MEASURES:

1. Primary Outcome: Summary of Number of Participants With Treatment Emergent Adverse Events (TEAE) - All Grades
Description: Adverse events (AEs), serious adverse events (SAEs), changes from baseline in vital signs and laboratory results (hematology, blood chemistry, lipid profile) qualifying and reported as AEs. Although a patient might had two or more adverse events the patient is only counted once in a category. The same patient might appear in different categories. AESI: Adverse events of special interest.
Time Frame: Baseline up to approximately 43 weeks for Asian countires and 32 weeks for Non-Asian countries including a 30 day post treatment follow up period
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Total: Asian and Non -Asian countries
Arm/Group | Asian Everolimus + Exemestane | Non-Asian Everolimus + Exemestane | Total
Number analyzed (Participants) | 199 | 36 | 235
Participants
  no TEAE | 4 | 0 | 4
  at least 1 TEAE | 195 | 36 | 231
  at least 1 drug-related TEAE | 185 | 33 | 218
  at least 1 serious TEAE (STEAE) | 59 | 16 | 75
  STEAE leading to death | 6 | 4 | 10
  Non-fatal STEAE | 53 | 12 | 65
  at least 1 drug-related STEAE | 28 | 8 | 36
  at least 1 drug-related STEAE - death | 2 | 1 | 3
  at least 1 drug-related non-fatal STEAE | 26 | 7 | 33
  TEAE leading to permanent tx discontinuation | 25 | 11 | 36
  1 TE AESI | 172 | 34 | 206

2. Secondary Outcome: Percentage of Participants Response Rates (Best Overall and Overall)
Description: The best overall response for each patient is determined from the sequence of investigator overall lesion responses according to RECIST 1.1: Complete Response (CR)=disappearance of target lesions, Partial Response (PR) was >=30% decrease in sum of diameter of lesions, Progressive Disease (PD) was >=20% decrease in sum of diameter of lesions, Stable Disease (SD) does not qualify for PR, CR or PD, Unknown=not documented or assessed. To be assigned a best overall response of CR at least two determinations of CR at least 4 weeks apart before progression are required. To be assigned a best overall response of PR at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) are required. The Overall response rate (ORR) is the percentage of patients with a best overall response of confirmed complete (CR) or partial (PR) response. The 95% confidence intervals (CI) were computed using the Clopper-Pearson method
Time Frame: Baseline up to approximately 43 weeks for Asian countires and 32 weeks for Non-Asian countries
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Total: Asian and Non-Asianb
Arm/Group | Asian Everolimus + Exemestane | Non-Asian Everolimus + Exemestane | Total
Number analyzed (Participants) | 199 | 36 | 235
Percentage of participants
  Complete response (CR) | 1.5 [0.3 to 4.3] | 0.00 [NA to NA] — Not available for 0 percent response | 1.3 [0.3 to 3.7]
  Partial response (PR) | 20.1 [14.8 to 26.3] | 8.3 [1.8 to 22.5] | 18.3 [13.6 to 23.8]
  Stable disease (SD) | 51.3 [44.1 to 58.4] | 63.9 [46.2 to 79.2] | 53.2 [46.6 to 59.7]
  Progressive disease (PD) | 18.1 [13.0 to 24.2] | 19.4 [8.2 to 36.0] | 18.3 [13.6 to 23.8]
  Unknown (UNK) | 9.0 [5.4 to 13.9] | 8.3 [1.8 to 22.5] | 8.9 [5.6 to 13.3]
  Overall response rate (ORR: CR+PR) | 21.6 [16.1 to 28.0] | 8.3 [1.8 to 22.5] | 19.6 [14.7 to 25.2]

3. Secondary Outcome: Percentage of Participants Clinical Benefit Rate
Description: Clinical benefit rate: Patients with best overall response rate of CR (any duration), PR (any duration) and SD with duration of 24 weeks or longer according to RECIST 1.1 criteria: Complete Response (CR)=disappearance of target lesions, Partial Response (PR) was >=30% decrease in sum of diameter of lesions, Progressive Disease (PD) was >=20% decrease in sum of diameter of lesions, Stable Disease (SD) does not qualify for PR, CR or PD, Unknown=not documented or assessed. Best overall response of CR = at least two determinations of CR at least 4 weeks apart before progression are required. Best overall response of PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) are required. The Overall response rate (ORR) is the percentage of patients with a best overall response of confirmed complete (CR) or partial (PR) response. The 95% confidence intervals (CI) were computed using the Clopper-Pearson method.
Time Frame: Baseline up to approximately 43 weeks for Asian countires and 32 weeks for Non-Asian countries
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Asian Everolimus + Exemestane | Non-Asian Everolimus + Exemestane | Total
Number analyzed (Participants) | 199 | 36 | 235
Percentage of participants | 48.2 [41.1 to 55.4] | 30.6 [16.3 to 48.1] | 45.5 [39.0 to 52.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is time from date of start of treatment to date of disease progression or death due to any cause, whichever occurs first.
  b Percentiles with 95% CIs are calculated from PROC LIFETEST output using method of Brookmeyer and Crowley (1982)
Time Frame: Baseline up to approximately 43 weeks for Asian countires and 40 weeks for Non-Asian countries
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Asian Everolimus and Exemestane: Everolimus (10 mg) and exemestane (25 mg) tablets taken orally in combination once daily. Participants in Asian countries: Indonesia, India, Vietnam, Turkey, South Korea, Thailand, Malaysia, Taiwan or Jordan
- Total: Asian and Non-Asian countries
Arm/Group | Asian Everolimus and Exemestane | Non-Asian Everolimus + Exemestane | Total
Number analyzed (Participants) | 199 | 36 | 235
weeks | 40.6 [39.3 to 50.3] | 37.0 [26.7 to 52.0] | 40.6 [38.0 to 48.9]

5. Secondary Outcome: Percent of Participants Event-free Probability Estimates of Deterioration of Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Time to deterioration of ECOG performance status, from baseline will be assessed using the ECOG Performance Status Scale (Oken, 1982). Time to deterioration is the time from date of start of treatment to the date of the event defined as deterioration. Deterioration is defined as an increase in performance status from 0 to 2 or greater, an increase in performance status from 1-2 to 3 or greater, or death due to any cause. Event-free probability estimate is the estimated probability that a patient will remain event-free up to the specified time point. Event-free probability estimates were are obtained from the Kaplan-Meier survival estimates.
Time Frame: Baseline up to approximately 50 weeks
Population: Number of participants meeting criteria differed at visits
Measure: Number; unit: percent of participants
Arm/Group | Asian Everolimus + Exemestane | Non-Asian Everolimus + Exemestane | Total
Number analyzed (Participants) | 199 | 36 | 235
percent of participants
  Week 0 n=199,36,235 | 100.0 | 100.0 | 100.00
  Week 20 n=134,18,152: number analyzed (Participants) | 134 | 18 | 152
  Week 20 n=134,18,152 | 95.0 | 79.8 | 92.7
  Week 50 n=58,7,65: number analyzed (Participants) | 58 | 7 | 65
  Week 50 n=58,7,65 | 90.6 | 70.4 | 87.6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration off approximately 43 weeks for Asian countries and 32 weeks for Non-Asian countries
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- Asian: Everolimus (10 mg) and exemestane (25 mg) tablets taken orally in combination once daily. Participants in Asian countries: Indonesia, India, Vietnam, Turkey, South Korea, Thailand, Malaysia, Taiwan or Jordan.
- Non-Asian: Everolimus (10 mg) and exemestane (25 mg) tablets taken orally in combination once daily. Participants in Non-Asian countries: Australia, Morocco, South Africa or Tunisia.
Arm/Group | Asian | Non-Asian
All-Cause Mortality (participants affected / at risk) | 6/199 | 4/36
Serious Adverse Events (participants affected / at risk) | 59/199 | 16/36
Other Adverse Events (participants affected / at risk) | 192/199 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asian (N=199) | Non-Asian (N=36)
Anaemia (Blood and lymphatic system disorders) | 7 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 2 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 3 | 1
Gait inability (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 5 | 3
Contrast media allergy (Immune system disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 2
Herpes virus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 1
Sepsis (Infections and infestations) | 0 | 2
Soft tissue infection (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Urosepsis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Eastern cooperative oncology group performance status worsened (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asian (N=199) | Non-Asian (N=36)
Anaemia (Blood and lymphatic system disorders) | 38 | 8
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 4
Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 10 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 12 | 3
Dental caries (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 30 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 15 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 1
Mouth ulceration (Gastrointestinal disorders) | 7 | 9
Nausea (Gastrointestinal disorders) | 23 | 9
Oral pain (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 125 | 14
Toothache (Gastrointestinal disorders) | 8 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4
Asthenia (General disorders) | 10 | 2
Face oedema (General disorders) | 5 | 0
Fatigue (General disorders) | 31 | 14
Influenza like illness (General disorders) | 4 | 0
Mucosal inflammation (General disorders) | 4 | 0
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 16 | 5
Pain (General disorders) | 3 | 2
Peripheral swelling (General disorders) | 8 | 1
Pyrexia (General disorders) | 12 | 3
Swelling (General disorders) | 0 | 1
Unevaluable event (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 5 | 1
Ear infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 2 | 1
Furuncle (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 6 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 6 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 10 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 23 | 2
Urinary tract infection (Infections and infestations) | 9 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 45 | 4
Aspartate aminotransferase increased (Investigations) | 50 | 3
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 9 | 1
Blood cholesterol increased (Investigations) | 32 | 4
Blood creatinine increased (Investigations) | 7 | 0
Blood lactate dehydrogenase increased (Investigations) | 17 | 2
Blood triglycerides increased (Investigations) | 4 | 0
Breath sounds abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 30 | 2
Haemoglobin decreased (Investigations) | 5 | 0
Liver function test abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Liver palpable (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 10 | 0
Platelet count decreased (Investigations) | 4 | 1
Weight decreased (Investigations) | 32 | 4
White blood cell count decreased (Investigations) | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 53 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 10 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 51 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 23 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 2
Dizziness postural (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 13 | 4
Headache (Nervous system disorders) | 23 | 4
Hypoaesthesia (Nervous system disorders) | 4 | 0
Paraesthesia (Nervous system disorders) | 5 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 5 | 0
Insomnia (Psychiatric disorders) | 18 | 5
Breast pain (Reproductive system and breast disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 4
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 25 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 8 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 3
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 2 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 4 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 2
Rash (Skin and subcutaneous tissue disorders) | 48 | 12
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 1
Hot flush (Vascular disorders) | 1 | 5
Hypertension (Vascular disorders) | 12 | 1
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 10 | 2
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT03176238/SAP_000.pdf
  • Study Protocol (2014-07-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT03176238/Prot_001.pdf